CLINICAL TRIAL: NCT06073951
Title: Mates in Motion: Feasibility and Acceptability of a Couple-Based Physical Activity Intervention
Brief Title: Evaluation of a Couple-Based Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-008130; NCI-2023-07197 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-008130 (Other: Mayo Clinic in Arizona); R21CA275085-01A1 (NIH)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Mates in Motion) (Experimental): Dyads participate in the Mates in Motion program consisting of weekly sessions to train couples in the use of communal coping strategies to support one another in achieving PA goals and skill building focus on instruction and practice in effective communication, with emphases on adaptive speaking, responsive listening, and joint decision-making and problem-solving around PA over 8 weeks. Patient-partner dyads receive weekly step-count goals, complete walk-tests and questionnaires and wear an Actigraph device and Garmin activity tracker on study.
  Interventions: Other: Exercise Counseling; Other: Exercise Intervention; Other: Medical Device Usage and Evaluation; Other: Physical Performance Testing; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patient-partner dyads wear an Actigraph device, compete walk-tests and questionnaires on study. Dyads receive usual care on study. Dyads receive a Garmin activity tracker at the end of the study.
  Interventions: Other: Best Practice; Other: Medical Device Usage and Evaluation; Other: Physical Performance Testing; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Other: Exercise Counseling — Receive walking step goals
  Arms: Arm I (Mates in Motion)
Other: Exercise Intervention — Participate in Mates in Motion program
  Arms: Arm I (Mates in Motion)
Other: Medical Device Usage and Evaluation — Wear Actigraph
  Arms: Arm I (Mates in Motion)
Other: Medical Device Usage and Evaluation — Wear Garmin activity tracker
Other: Physical Performance Testing — Undergo walk-test
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial tests how well a couple-based physical activity (PA) intervention, Mates in Motion, works in patients undergoing hematopoietic cell transplantation (HCT) or chimeric antigen receptor T-cell therapy (CART) and their care giving partners to be more physically active. Mates in Motion provides training in communication skills and behavior change techniques to help HCT patient-caregiver dyads support one another in adoption and maintenance of PA. This study may help researchers determine if a couple-based PA intervention improves PA, physical endurance and global physical health among patient-care giver dyads undergoing HCT or CART.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine feasibility of recruitment, adherence, and retention of a couple-based PA intervention in a pilot randomized controlled trial (RCT).

II. Determine acceptability of the intervention (multiple dimensions of treatment satisfaction).

III. Describe changes in PA, physical endurance, and global physical health from baseline to follow-up as a function of randomized condition.

OUTLINE: Patient-caregiver dyads are randomized to 1 of 2 arms.

ARM I: Dyads participate in the Mates in Motion program consisting of weekly sessions to train couples in the use of communal coping strategies to support one another in achieving PA goals and skill building focus on instruction and practice in effective communication, with emphases on adaptive speaking, responsive listening, and joint decision-making and problem-solving around PA over 8 weeks. Patient-partner dyads receive weekly step-count goals, complete walk-tests and questionnaires and wear an Actigraph device and Garmin activity tracker on study.

ARM II: Patient-partner dyads wear an Actigraph device, compete walk-tests and questionnaires on study. Dyads receive usual care on study. Dyads receive a Garmin activity tracker at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Age 18 years or older
* PATIENTS: Scheduled to receive an autologous or allogeneic hematopoietic cell transplant (HCT) or chimeric antigen receptor (CAR)-T cell therapy
* PATIENTS: Able to speak and comprehend English
* PATIENTS: Being married or in a committed (self-defined) cohabiting same- or opposite-sex relationship
* PATIENTS: Physician-approved for a walking program
* CAREGIVERS: Age 18 years or older
* CAREGIVERS: Able to speak and comprehend English
* CAREGIVERS: Married to or in a committed, cohabiting, same- or opposite-sex relationship with the patient
* CAREGIVERS: Able to participate in a walking program

Exclusion Criteria:

* None per se beyond the converse of the inclusions listed above, for example, age younger than 18 years and non-partnered

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Observed recruitment | At baseline
  Will be assessed by the percentage of eligible patient-partner couples agreeing to participate
Intervention adherence | 8 weeks
  Will be assessed by the number of intervention sessions attended.
Actigraph wear adherence | 8 weeks
  Will be assessed by the number of valid wear days.
Garmin wear adherence | 8 weeks
  Will be assessed by the number of valid wear days.
Retention | At 100 days post-hematopoietic cell transplant (HCT)
  Will be assessed by the number of post-intervention follow-up assessments completed.

SECONDARY OUTCOMES:
Acceptability of the intervention | At 100 days post-hematopoietic cell transplant (HCT)
  Will be assessed among patients and caregivers and will examine ratings for the following treatment satisfaction domains relative to the scale midpoint: suitability, utility, attitude toward treatment, desire for continued treatment use, therapist competence, therapist interpersonal style, format and dose, and perceived benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Nandita Khera, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT06073951/ICF_000.pdf